CLINICAL TRIAL: NCT03687749
Title: Presentation of First Time Attenders at Lymphedema Clinics: Cross-sectional Study
Brief Title: Presentation of First Time Attenders at Lymphedema Clinics
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Sponsor
Other Study IDs: S59883
Record Dates: First submitted 2018-07-10; First posted 2018-09-27 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Lymphedema; Breast Neoplasm
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with breast cancer-related lymphedema: Individuals with upper limb lymphedema developed after breast cancer treatment
- Healthy control subjects: Healthy individuals without breast cancer-related lymphoedema.

SUMMARY:
The first aim of this research project is to identify what factors motivate patients to seek assessment for early lymphedema and further, to gain insight into the signs and symptoms of developing lymphedema and the concurrent physical measurements.

The second aim is to identify other sensory signs and symptoms and changes in body perception which may be perceived by the patient as reflective of lymphedema, and to identify to which degree they contribute to the patients' motivation to seek referral to lymphedema clinics.

DETAILED DESCRIPTION:
One of the most challenging morbidities after breast cancer treatment is lymphedema. Approximately 20% of women treated for breast cancer with axillary lymph node dissection will be diagnosed with lymphedema. Pre- and post-operatively, women are informed about changes suggestive of lymphedema and guided about seeking further assessment. The investigators presume that if symptoms occur, patients will seek assessment. However, it is unknown whether this is true or if those prospectively monitored present earlier for treatment, or whether other factors specifically drive patients to seek further assessment. Understanding the early experience and presentation of secondary lymphedema will improve patient education and detection programs.

ELIGIBILITY:
Inclusion Criteria:

* women after breast cancer (> 18 years) with unilateral axillary lymph node dissection or sentinel node biopsy; mastectomy (with or without autologous reconstruction) or wide excision of the tumor
* able to give consent to participate in the research

Exclusion Criteria:

* patients under the age of 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two hundred women who have previously been treated for unilateral breast cancer and are referred for the first time to a lymphedema clinic. These patients presenting for the first time with breast cancer-related lymphedema will be asked to have an immediate objective assessment of their lymphedema and to administer additional questionnaires and clinical tests.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Extracellular fluid in the arm | immediately after inclusion in the study
  Bioimpedance spectroscopy (BIS) is a measurement tool used to determine the volume of extracellular fluid, of which lymph fluid is a component.
Arm volume | immediately after inclusion in the study
  Arm circumference measures are commonly used to diagnose and monitor lymphedema.
Pitting | immediately after inclusion in the study
  The pitting tests examines the responsiveness of tissue to pressure and can be used to help determine the stage of lymphedema.

SECONDARY OUTCOMES:
Self-reported signs and symptoms of lymphedema | immediately after inclusion in the study
  Norman questionnaire for early detection of lymphedema will be used; this validated questionnaire will allow us to determine the location and severity of the symptoms that the patients have experienced over the past three months as well as how much distress it has caused.
Impairments in function, activity limitations, and participation restrictions of patients with arm lymphedema | immediately after inclusion in the study
  Lymphoedema Functioning, Disability and Health questionnaire (Lymph-ICF): The Lymph-ICF is a reliable and valid questionnaire to assess impairments in function, activity limitations, and participation restrictions of patients with arm lymphedema.
Global Health Status/Quality of Life Score | immediately after inclusion in the study
  Health-related quality of life assessed with the generic QLQ-C30 and the disease-specific QLQ-BR23 questionnaire
Body perception | immediately after inclusion in the study
  The BATH CRPS body perception disturbances scale: to assess body perception disturbances in breast cancer patients.
Pain intensity assessed with the Numeric Rating Scale | immediately after inclusion in the study
  Numeric Rating Scale for maximal pain intensity during the past week.
Prevalence of neuropathic pain | immediately after inclusion in the study
  Measured with the Douleur Neuropathique en 4 questions (DN4)
Tactile acuity (Two-point discrimination) | immediately after inclusion in the study
  To assess body perception two-point discrimination will be assessed at both arms, the breasts and lateral trunk side.
Mechanical detection and pain threshold | immediately after inclusion in the study
  The lowest mechanical forces, applied to the skin using nylon monofilaments that the subject can 1) detect and 2) is perceived as painful) are tested at the upper limb and upper body region.
Temporal summation | immediately after inclusion in the study
  Detection of perceived temporal summation at the upper limb and upper body region tested using repeated 26g nylon monofilament stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: An De Groef, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Elizabeth Dylke, PhD, Principal Investigator — University of Sydney, Faculty of Health Sciences
Locations (2):
- University of Sydney, Faculty of Health Sciences, Sydney, New South Wales, Australia
- University Hospital Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No